CLINICAL TRIAL: NCT07395349
Title: Safety And Recovery Of Tubeless Strategy In Uniportal VATS Wedge Resection: A Single-Center, Prospective Randomized Controlled Study Based On Different Intraoperative Pleural Space Management Strategies
Brief Title: Safety And Recovery Of Tubeless Strategy In Uniportal VATS Wedge Resection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, Department of Thoracic Surgery, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GYFYY-THOR-TUBELESS-RCT-2026-0
Record Dates: First submitted 2026-01-25; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Nodule; Pneumothorax; Postoperative Complications
Keywords: Uniportal VATS; Wedge Resection; Tubeless; Intraoperative Aspiration; Chest Tube Drainage; Enhanced Recovery After Surgery (ERAS); Lung Re-expansion
MeSH Terms: conditions — Pneumothorax; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Participants who meet intraoperative eligibility criteria are randomized in a 1:1:1 ratio to three parallel groups receiving different intraoperative pleural space management strategies.
Masking Description: This is an open-label surgical trial. Due to the nature of the interventions, masking of participants, care providers, and investigators is not feasible. Outcome assessments are based on objective clinical events and standardized evaluation criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Chest Tube Drainage (CTD) (Active Comparator): Participants undergo uniportal VATS wedge resection followed by routine postoperative chest tube drainage. A chest tube is placed at the end of surgery and managed according to standard institutional protocols, including water seal or suction, criteria for tube removal, and discharge standards. This arm serves as the control group for comparison with tubeless strategies.
  Interventions: Procedure: Conventional Chest Tube Drainage
- Single Intraoperative Aspiration Tubeless (SIA-Tubeless) (Experimental): Participants undergo uniportal VATS wedge resection and, after passing a standardized intraoperative water-seal air leak test, receive a single intraoperative negative-pressure aspiration of the pleural space under positive-pressure ventilation before chest closure. The catheter is completely removed intraoperatively, and no postoperative chest tube or aspiration is permitted.
  Interventions: Procedure: Single Intraoperative Aspiration Tubeless
- Double Intraoperative Aspiration Tubeless (DIA-Tubeless) (Experimental): Participants undergo uniportal VATS wedge resection and, after passing a standardized intraoperative water-seal air leak test, receive two consecutive intraoperative negative-pressure aspirations of the pleural space under positive-pressure ventilation before chest closure. After the second aspiration, the catheter is completely removed. No postoperative chest tube or aspiration is permitted.
  Interventions: Procedure: Double Intraoperative Aspiration Tubeless

INTERVENTIONS:
Procedure: Conventional Chest Tube Drainage — After uniportal VATS wedge resection, a chest tube is routinely placed at the end of surgery for postoperative pleural drainage. Chest tube management, including water seal or suction, criteria for tube removal, and discharge standards, follows standard institutional protocols.
  Other Names: CTD
  Arms: Conventional Chest Tube Drainage (CTD)
Procedure: Single Intraoperative Aspiration Tubeless — After uniportal VATS wedge resection and confirmation of no persistent air leak using a standardized intraoperative water-seal air leak test, a single negative-pressure aspiration of the pleural space is performed intraoperatively under positive-pressure ventilation before chest closure. The aspiration catheter is completely removed intraoperatively, and no postoperative chest tube or aspiration is allowed.
  Other Names: SIA-Tubeless
  Arms: Single Intraoperative Aspiration Tubeless (SIA-Tubeless)
Procedure: Double Intraoperative Aspiration Tubeless — After uniportal VATS wedge resection and confirmation of no persistent air leak using a standardized intraoperative water-seal air leak test, two consecutive negative-pressure aspirations of the pleural space are performed intraoperatively under positive-pressure ventilation before chest closure. After the second aspiration, the catheter is completely removed. No postoperative chest tube or aspiration is permitted.
  Other Names: DIA-Tubeless
  Arms: Double Intraoperative Aspiration Tubeless (DIA-Tubeless)

SUMMARY:
Brief Summary

The goal of this clinical trial is to evaluate the safety and recovery outcomes of different tubeless strategies in adult patients undergoing uniportal video-assisted thoracoscopic (VATS) wedge resection who are confirmed to have no persistent air leak intraoperatively.

The main questions it aims to answer are:

Does double intraoperative aspiration tubeless strategy reduce the rate of postoperative pleural re-intervention within 30 days compared with single intraoperative aspiration tubeless strategy?

Do different intraoperative pleural space management strategies affect early postoperative recovery quality and pain?

If there is a comparison group:

Researchers will compare conventional chest tube drainage, single intraoperative aspiration tubeless, and double intraoperative aspiration tubeless strategies to determine their effects on postoperative pleural re-intervention and recovery outcomes.

Participants will:

Undergo uniportal VATS wedge resection

Receive a standardized intraoperative air leak test before chest closure

Be randomly assigned intraoperatively to one of three pleural space management strategies

Complete postoperative assessments including chest imaging, pain evaluation, and recovery quality questionnaires

Be followed for 30 days after surgery for safety outcomes

DETAILED DESCRIPTION:
Uniportal video-assisted thoracoscopic (VATS) wedge resection is widely used for the diagnosis and treatment of peripheral pulmonary nodules. Conventional postoperative chest tube drainage is routinely applied to prevent pneumothorax, but it is associated with increased postoperative pain, delayed mobilization, and prolonged hospital stay. In recent years, tubeless strategies have been introduced in carefully selected patients to enhance recovery; however, postoperative residual pneumothorax and pleural re-intervention remain major safety concerns.

Previous retrospective studies suggest that intraoperative aspiration may improve the feasibility of tubeless VATS, but single aspiration may not completely prevent re-entry of air into the pleural space. A modified strategy using double intraoperative aspiration performed entirely before chest closure may enhance lung re-expansion and reduce postoperative pleural complications. To date, no prospective randomized controlled trial has directly compared different intraoperative aspiration-based tubeless strategies.

This study is a single-center, prospective, three-arm randomized controlled trial conducted at Guangzhou Medical University First Affiliated Hospital. Adult patients undergoing uniportal VATS wedge resection who pass a standardized intraoperative water-seal air leak test will be randomized in a 1:1:1 ratio to one of the following groups:

conventional chest tube drainage,

single intraoperative aspiration tubeless, or

double intraoperative aspiration tubeless.

All aspiration procedures are completed intraoperatively, and no postoperative aspiration or intermittent drainage is permitted in tubeless groups. Perioperative management is standardized across all groups.

The primary outcome is the incidence of pleural re-intervention (thoracentesis or chest tube insertion) within 30 days after surgery. Secondary outcomes include postoperative recovery quality assessed by the QoR-15 questionnaire, postoperative pain assessed by visual analog scale (VAS), lung re-expansion on postoperative day 1 imaging, length of hospital stay, and postoperative pulmonary complications.

This trial aims to provide high-quality evidence to determine whether optimization of intraoperative pleural space management can improve the safety and reliability of tubeless uniportal VATS wedge resection while preserving enhanced recovery benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years
2. Scheduled to undergo uniportal video-assisted thoracoscopic (VATS) wedge resection
3. Able to tolerate general anesthesia and single-lung ventilation
4. Passed a standardized intraoperative water-seal air leak test, confirming absence of persistent air leak before chest closure
5. Able and willing to provide written informed consent
6. Able to complete postoperative assessments and 30-day follow-up

Exclusion Criteria:

1. Planned anatomical lung resection (segmentectomy or lobectomy) or combined complex thoracic procedures
2. Extensive pleural adhesions, severe emphysema, bullous lung disease, or other conditions associated with high risk of air leak
3. Positive intraoperative air leak test indicating persistent air leak
4. Requirement for additional intraoperative procedures that may significantly affect pleural air leak or lung re-expansion
5. Conversion to multiport VATS or thoracotomy before randomization
6. Severe comorbidities or other conditions deemed by the investigators to make participation inappropriate
7. Inability to complete follow-up or insufficient clinical data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Pleural Re-intervention Within 30 Days | From surgery to 30 days postoperatively
  Incidence of pleural re-intervention within 30 days after surgery, defined as thoracentesis or chest tube insertion performed for postoperative pneumothorax or residual intrapleural air.

SECONDARY OUTCOMES:
Lung Re-expansion on Postoperative Day 1 Chest X-ray | Postoperative day 1
  Residual pneumothorax / lung re-expansion status assessed on postoperative day 1 chest X-ray using a predefined grading or qualitative evaluation.
Postoperative Pain (VAS) Score | Postoperative day 1 and at hospital discharge, assessed up to 30 days after surgery
  Pain intensity assessed using a Visual Analog Scale (VAS), range 0-10, where higher scores indicate more severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of GZMU, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcome results, including baseline characteristics, intervention assignment, and outcome measures, will be shared.
Supporting Information: Study Protocol
Time Frame: IPD and supporting information will be available after publication of the primary study results, beginning approximately 6 months after publication, and will remain available for up to 5 years.
Access Criteria: Access to de-identified IPD and supporting information will be granted to qualified researchers upon reasonable request. Requests must include a brief research proposal and analysis plan and be approved by the study investigators. Data will be shared for academic research purposes only, without any attempt to re-identify participants. Data will be provided through secure data transfer methods.

REFERENCES:
- [Result] Yang Q, Lv S, Li Q, Lan L, Sun X, Feng X, Han K. Safety and feasibility study of uniportal video-assisted thoracoscopic pulmonary wedge resection without postoperative chest tube drainage: a retrospective propensity score-matched study. Interdiscip Cardiovasc Thorac Surg. 2022 Jan 1;37(6):ivad196. doi: 10.1093/icvts/ivad196. PMID 38092062
- [Result] Ueda K, Haruki T, Murakami J, Tanaka T, Hayashi M, Hamano K. No Drain After Thoracoscopic Major Lung Resection for Cancer Helps Preserve the Physical Function. Ann Thorac Surg. 2019 Aug;108(2):399-404. doi: 10.1016/j.athoracsur.2019.03.018. Epub 2019 Apr 5. PMID 30959014
- [Result] Batchelor TJP, Rasburn NJ, Abdelnour-Berchtold E, Brunelli A, Cerfolio RJ, Gonzalez M, Ljungqvist O, Petersen RH, Popescu WM, Slinger PD, Naidu B. Guidelines for enhanced recovery after lung surgery: recommendations of the Enhanced Recovery After Surgery (ERAS(R)) Society and the European Society of Thoracic Surgeons (ESTS). Eur J Cardiothorac Surg. 2019 Jan 1;55(1):91-115. doi: 10.1093/ejcts/ezy301. PMID 30304509
- [Result] Yang SM, Wang ML, Hung MH, Hsu HH, Cheng YJ, Chen JS. Tubeless Uniportal Thoracoscopic Wedge Resection for Peripheral Lung Nodules. Ann Thorac Surg. 2017 Feb;103(2):462-468. doi: 10.1016/j.athoracsur.2016.09.006. Epub 2016 Nov 16. PMID 27865474